CLINICAL TRIAL: NCT06789276
Title: The Impact of Thoracic Paravertebral Nerve Block At Different Positions on Pain Relief in Patients Undergoing Single-Port Thoracoscopic Partial Lung Resection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JD-LK2023067-I01
Record Dates: First submitted 2025-01-10; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Lung Nodules; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Supine Position

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- supine group (Experimental): This study selected patients scheduled for thoracoscopic lung resection at the Second Affiliated Hospital of Soochow University. The patients were divided into two groups using a random number table: the supine group and the lateral decubitus group. Patients who are placed in the supine position after the intervention are assigned to the supine group.
  Interventions: Behavioral: Supine position
- lateral decubitus group (Experimental): This study selected patients scheduled for thoracoscopic lung resection at the Second Affiliated Hospital of Soochow University. The patients were divided into two groups using a random number table: the supine group and the lateral decubitus group. Patients who are placed in the lateral decubitus position on the affected side after the intervention are assigned to the lateral decubitus group.
  Interventions: Behavioral: lateral decubitus position

INTERVENTIONS:
Behavioral: Supine position — For patients scheduled for thoracoscopic surgery, thoracic paravertebral nerve block was performed under ultrasound guidance. After the injection of the drug, patients were positioned in either the supine position.
  Arms: supine group
Behavioral: lateral decubitus position — For patients scheduled for thoracoscopic surgery, thoracic paravertebral nerve block was performed under ultrasound guidance. After the injection of the drug, patients were positioned in the lateral decubitus position with the puncture side up.
  Arms: lateral decubitus group

SUMMARY:
Thoracic surgery is widely recognized as one of the most painful surgical procedures. Compared to open thoracotomy, video-assisted thoracoscopic surgery (VATS) offers similar therapeutic outcomes with less invasiveness, significantly reducing postoperative pain and promoting recovery. Despite the use of video-assisted thoracoscopic surgery (VATS), a significant proportion of patients still experience considerable discomfort. Specifically, 78% of patients report moderate to severe pain, with 27% experiencing moderate pain, 34% severe pain, and 17% very severe pain.

Multiple studies have shown that the use of regional anesthesia, such as thoracic paravertebral nerve block (TPVB), in these surgeries can block the transmission of nociceptive signals via the intercostal nerves, producing good analgesic effects. This can reduce the consumption of postoperative opioids, decrease inflammatory responses, and improve patient survival rates after surgery.

By comparing the differences in hemodynamic parameters, inflammatory stress indicators, and intraoperative and postoperative analgesic effects of thoracic paravertebral nerve block in different preoperative positions for patients undergoing thoracoscopic surgery, we aim to identify the optimal nerve block position, thereby promoting patient recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 70 years old

  * BMI ≥ 18 and ≤ 28

    * American Society of Anesthesiologists (ASA) physical status classification I-II ⑷ Patients scheduled for elective thoracoscopic lung resection (including lobectomy, segmentectomy, and wedge resection) ⑸ Patients who agree to participate in this study and sign the informed consent form

Exclusion Criteria:

* Patients who refuse to undergo nerve block

  * Patients with severe cardiac, pulmonary, hepatic, or renal insufficiency requiring postoperative admission to the ICU for continued treatment (EF < 40%, FEV1/FVC < 40%)

    * Abnormal coagulation function ⑷ History of allergy to anesthetic drugs

      * History of chronic alcohol use, chronic pain, or long-term use of psychotropic medications ⑹ Scars, infections, or tumors at the puncture site ⑺ History or family history of malignant hyperthermia ⑻ Refusal to participate in this study or inability to cooperate with follow-up or poor compliance

Termination criteria:

* Failure to comply with the predetermined study protocol ⑵ Occurrence of local anesthetic adverse reactions, puncture needle entering the pleural cavity, or other complications during puncture

  * Changes in the patient's condition ⑷ The patient's unwillingness to continue participating in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-18 (Estimated); Primary Completion 2025-08-07 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Using the Numeric Rating Scale (NRS) scores to assess the postoperative analgesic effect in patients | For each patient enrolled in the study, data collection will commence at the time of enrollment and continue through to 48 hours postoperatively. The timeframe for conducting data analysis and reporting will be capped at one year.
  The primary outcome is to assess the patients' pain levels at 1h, 2h, 8h, 12h, 24h, and 48h postoperatively, as well as the analgesic efficacy of the nerve block, using the Numeric Rating Scale (NRS) scores for static (lying or sitting) and dynamic (coughing) conditions.
  The Numeric Rating Scale (NRS) is a simple and effective tool for assessing the intensity of pain, widely used in clinical settings and research. The NRS score is determined by asking patients to select a number between 0 and 10 to represent their level of pain, where 0 indicates no pain and 10 indicates the most severe pain. Specifically, 0 represents no pain, 1-3 represents mild pain, 4-6 represents moderate pain, and 7-10 represents severe pain.

SECONDARY OUTCOMES:
Using the postoperative opioid consumption to assess the postoperative analgesic effect in patients. | For each enrolled patient,data collection will commence at the time of enrollment and continue through to 24 hours postoperatively. The period for data analysis and reporting will not exceed one year.
  The secondary outcome is to assess the total amount of opioids (such as sufentanil) used by patients within 24 hours postoperatively.
  By comparing the opioid consumption between two groups of patients, it is possible to determine which treatment plan is more effective in controlling postoperative pain. The amount of opioid consumption can indirectly reflect the postoperative recovery status of patients. Lower consumption generally indicates better pain control and better recovery. Reducing the use of opioids can decrease the incidence of adverse reactions such as postoperative nausea, vomiting, and respiratory depression, thereby improving the postoperative quality of life of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zhu X, Peng P, Guo J, Zhang L, Zhong H, Zhu J, Xie H. The impact of thoracic paravertebral nerve block at different positions on pain relief in patients undergoing single-port thoracoscopic partial lung resection: study protocol for a randomized controlled trial. Trials. 2026 Feb 3;27(1):99. doi: 10.1186/s13063-025-09198-7. PMID 41634718